CLINICAL TRIAL: NCT03317470
Title: Addressing Unmet Basic Needs to Improve Adherence Among Women With an Abnormal Pap
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 201708116
Record Dates: First submitted 2017-10-09; First posted 2017-10-23 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Abnormal Pap Smear; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I: (Active Comparator): * In Phase 1 of the study (first five months), the investigators will enroll new patients when they call them to remind them of their first colposcopy appointment. If patients consent, the investigators also will assess their basic needs during the call. Those who screen positive for at least one unmet basic need, will be referred to the 2-1-1 helpline at their clinic visit (or this information will be sent to them if they miss their clinic visit).
  * All women enrolled in our study will be asked to complete our basic needs survey and take a follow-up survey at the time of their first colposcopy visit.
  * For patients in phase 1, the follow-up survey will only assess acceptability of the basic needs survey (five questions)
  Interventions: Other: Basic needs survey; Other: Follow-up survey
- Phase 2: (Experimental): -In Phase 2 of the study (second five months), new colposcopy patients will be approached and consented in a similar fashion as in Phase 1 and asked to complete the basic needs survey. However, this time, patients who screen positive with at least one unmet basic need will be offered assistance by a life navigator (a trained case manager) who will contact the patients by phone within 2 business days of completing the survey.
  The life navigator will connect patients with community resources in each area to help with their unmet basic needs.
  * All women enrolled in our study will be asked to complete our basic needs survey and take a follow-up survey at the time of their first colposcopy visit.
  * Patients enrolled in phase 2 will be asked the same five questions in addition to seven more assessing perceived effectiveness of the life navigator
  Interventions: Other: Basic needs survey; Behavioral: Life Navigator; Other: Follow-up survey; Other: Follow-up survey (phase II participants only)

INTERVENTIONS:
Other: Basic needs survey — -11 questions about food security, housing personal safety, neighborhood safety, childcare, and transportation
Behavioral: Life Navigator — * The life navigator will contact women identified with unmet basic needs within two business days of completing the baseline survey.
  * The life navigator in our study will: (1) identify and assess women's needs; (2) jointly generate solutions to address the needs; (3) develop plans to carry out the solutions, including; (4) help prioritize among multiple needs; (5) identify community resources that could help solve the problem; (6) determine eligibility for services; (7) help women access available resources by scheduling appointments and provide appointment reminders; (8) prepare women to interact with service agencies and/or act as an advocate on their behalf; (9) provide instrumental support such as arranging transportation; (10) actively intervene to resolve barriers to basic needs solutions; (11) oversee follow-up of problem solving actions; and (12) review progress made towards resolving unmet basic needs and adapt solutions accordingly.
  Arms: Phase 2:
Other: Follow-up survey — -5 questions about the acceptability of the basic needs survey
Other: Follow-up survey (phase II participants only) — -7 questions about the effectiveness of the life navigator
  Arms: Phase 2:

SUMMARY:
The investigators aim to improve adherence to follow-up recommendations for an abnormal Pap and effectively reduce disparities in cervical cancer risk and disease among rural and low-income urban women.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patients to colposcopy clinic at SIUM and WUSM
* Aged 18 years or older
* English speaking
* Able to provide verbal consent
* Diagnosis of abnormal pap will be confirmed by pathology report
* Member of all races and ethnic groups

Exclusion Criteria:

* Male
* Established colposcopy clinic patients
* Known diagnosis of cancer
* Pregnancy
* Incarcerated
* Unable to consent
* No access to a working contact phone number

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2018-12-09 (Actual)

PRIMARY OUTCOMES:
Participant adherence to initial colposcopy visit | At the time of initial colposcopy visit
  -Will use weekly clinic schedules to track adherence rates

SECONDARY OUTCOMES:
Number of unmet basic needs | -2 weeks prior to initial colposcopy visits
  -Data obtained from Basic Needs Survey
Type of unmet basic needs | -2 weeks prior to initial colposcopy visits
  -Data obtained from Basic Needs Survey
Participant adherence to recommended follow-up after initial colposcopy visit | At the time of initial colposcopy visit
  -Data will be collected for each participant to notate whether participant showed up for recommended follow-up visit and will be tabulated for all participants
Participant acceptability of the unmet basic needs survey | At the time of initial colposcopy visit
Participant perception of effectiveness of life navigator to assist with their unmet basic needs | At the time of initial colposcopy visit
  * Data collected on the follow-up survey
  * 7 questions asking the following
    * Was the patient navigator helpful (yes with comments/no)
    * What could the navigator done better (multiple choice and area to add comments)
    * Did you use any of the resources the navigator told you about (yes with comments/no)
    * Would you recommend this type of helper to a family member or friend (yes/no)
    * Were there parts you didn't like or didn't find helpful (yes with comments/no)
    * Do you think the patient navigator helped you get to your clinic appointments (yes/no)
    * If available, would you find it helpful to talk to the patient navigator more (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M Kuroki, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuroki L, Massad LS, Martin A, Liu J, Brown D, Leon A, Groesch K, Wilson T, Zeino Y, Diaz-Sylvester P, Delfino K, Hyon K, Kreuter M. Addressing Unmet Basic Needs to Improve Colposcopy Adherence Among Women With Abnormal Cervical Cancer Screening. J Low Genit Tract Dis. 2021 Apr 1;25(2):106-112. doi: 10.1097/LGT.0000000000000593. PMID 33631781
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu